CLINICAL TRIAL: NCT01441713
Title: Treatment Frequency and Satisfaction in Patients With Advanced Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Other Study IDs: HeH.750.19-25
Record Dates: First submitted 2011-09-09; First posted 2011-09-28 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Prostatic Neoplasms
Keywords: Hormone treatment; castration; Orchiectomy; treatment frequency; treatment satisfaction; side effects
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pharmaceutical group: Patients in pharmaceutical castration treatment for advanced prostate cancer
- Surgical group: Patients having undergone surgical castration treatment for advanced prostate cancer

SUMMARY:
Patients with advanced prostate cancer usually receive some kind of pharmaceutical castration or undergo surgical castration. At the investigators department the pharmaceutical treatment is most often given with a 3 month interval.

Over the last few years new drugs, which allow for lees frequent treatment, have been developed. The purpose of this study is to assess how the treatment affects patients and if our current patients would prefer to receive treatment at different intervals than they do at the present time. At the same time the investigators will assess how surgical treatment affects our patients. This will be assessed by patient questionnaires administered at our clinic.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of advanced prostate cancer
* Receiving hormone manipulation treatment (pharmaceutical castration) OR having undergone surgical castration (orchiectomy)

Exclusion Criteria:

* Inability to read/write Danish

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who are receiving pharmaceutical castration treatment (hormone treatment) at Herlev Hospital for advanced prostate cancer and men who have undergone surgical castration (Orchiectomy) and are in clinical control at Herlev Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Preferred treatment/control frequency for patients with advanced prostate cancer | Up to 1 year
  Preferred treatment frequency is assessed by patient answers to the question:
  "If treatments were equally effective from a medical standpoint - How often would you then prefer to receive treatment"

SECONDARY OUTCOMES:
Treatment satisfaction | Up to 1 year
  Treatment satisfaction ranging from "Very satisfied" til "Very unsatisfied" assessed by patient answers to the questionnaire
Side effects to treatment | Up to 1 year
  Side effects to treatment assessed by patient answers to the questionnaire
Treatment satisfaction, preferred frequency of clinical control, and side effects after surgical castration | Up to 1 year
  As a secondary endpoint the investigators will look at answers to satisfaction, wishes for control visits and side effects in the group of patients who received surgical castration for their advanced prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Fode, MD, Principal Investigator — Herlev Hospital, University of Copenhagen
Locations (1):
- Department of urology, Herlev Hospital, Herlev, Denmark